CLINICAL TRIAL: NCT07229352
Title: Mobility Performance in Daily Activities Among Children Wearing Single Vision and Myopia Control Spectacle Lenses
Brief Title: Mobility Performance in Daily Activities Among Children Wearing Spectacle Lenses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPRO-2507-001
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Myopia Progression; Juvenile Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SightGlass Vision Test Arm 1 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Novel spectacle lens design
- SightGlass Vision Test Arm 2 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Spectacle lenses

INTERVENTIONS:
Device: Novel spectacle lens design — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: SightGlass Vision Test Arm 1
Device: Spectacle lenses — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: SightGlass Vision Test Arm 2

SUMMARY:
The aim of this study is evaluate and compare the mobility performance of children in daily activities while wearing single vision spectacle lenses (control) versus myopia control spectacle lenses (test).

ELIGIBILITY:
Inclusion Criteria:

A participant is eligible for inclusion in the study if they meet the following criteria:

* Are between the ages of 6 and 12 years of age (inclusive) at the time of informed consent/assent.
* Can achieve a corrected visual acuity of 20/20 best-corrected (or equivalent logMAR).
* Have undergone a self-reported oculo-visual examination within the past two years.
* Have no active ocular disease.
* Are willing and able to adhere to instructions, study procedures, and maintain the appointment schedule.
* Have not previously worn or participated in myopia control contact lenses for more than one month and are not currently undergoing any form of myopia control treatment.
* The subject's parent(s) or legal guardian(s) must read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form.

Exclusion Criteria:

A participant will be excluded from the study if they meet any of the following conditions:

* Have any systemic disease that affects ocular health.
* Are currently using or have used, within the past 7 days, any systemic or topical medications that may impact ocular health.
* Are currently using or have used any topical ophthalmic agents with anti-muscarinic properties within 7 days prior to enrollment or at any point during the study. This includes, but is not limited to, atropine, scopolamine, pirenzepine, tropicamide, cyclopentolate, and homatropine.
* Have used any oral agents with anti-muscarinic properties for a chronic period (2 months or more) or short-term (within 7 days prior to enrollment). This includes, but is not limited to, gastrointestinal anti-spasmodic medications containing atropine, hyoscyamine, and dicyclomine.
* Have known developmental delays.
* Have participated in another clinical study in the last 7 days

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Reaction time: the time elapsed between the appearance or activation of a visual stimulus and the initiation of the participant's physical response | 2 months
Movement time: the time taken to complete the motor response after it has been initiated. | 2 months
Response accuracy: the correctness of the participant's response to each visual stimulus, measured by the number or percentage of correctly identified or responded-to stimuli. | 2 months

SECONDARY OUTCOMES:
Gait cycle events, such as initial foot contact with the ground and toe-off. It will be used to assess whether the type of eyewear affects natural gait patterns or mobility during peripheral vision tasks. | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern University Arizona College of Optometry, Glendale, Arizona, United States